CLINICAL TRIAL: NCT02164838
Title: A Phase 1 Study of the VEGF Receptor Tyrosine Kinase Inhibitor Axitinib (INLYTA, IND# TBD) in Children With Recurrent or Refractory Solid Tumors
Brief Title: VEGF Receptor Tyrosine Kinase Inhibitor Axitinib in Children With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1315
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Refractory or Recurrent Solid Tumors, Excluding CNS Tumors
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental)
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib
  Other Names: AG-013736, INLYTA®

SUMMARY:
This trial will be the first study of axitinib in children and adolescents. The primary objective of this Phase 1 trial is to determine a maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of axitinib in pediatric patients with refractory solid tumors. Additional objectives include measurement of pharmacokinetic and pharmacodynamic parameters, description of the toxicity profile of this agent in children and adolescents, and assessment of response within the confines of a Phase 1 trial. A standard rolling 6 design will be used for dose escalation. Further development of axitinib will focus on development of a joint cooperative group (COG/ECOG) Phase 2 study of axitinib in pediatric, adolescent and young adult translocation renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria

* Age: Patients must be > than 12 months and < 18 years of age at the time of study enrollment.
* Body Surface Area: Patients must have a BSA of ≥ 0.53 m2 at the time of study enrollment.
* Diagnosis: Patients with refractory or recurrent solid tumors (excluding CNS tumors) and patients with unresectable translocation positive renal cell carcinoma (tRCC) are eligible. Patients must have had histologic verification of malignancy at original diagnosis or relapse.
* The diagnosis of translocation morphology or TFE renal cell carcinoma is established by having characteristic morphology AND either a) strong nuclear TFE3 or TFEb staining on immunohistochemistry OR b) cytogenetic studies of the tumor demonstrating a TFE translocation OR c) fluorescent in situ hybridization (FISH) demonstrating a TFE translocation.
* Disease Status: Patients must have either measurable or evaluable disease
* Therapeutic Options: Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age . Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy
* Patients may have received bevacizumab, VEGF-Trap, or other VEGF blocking tyrosine kinase inhibitors, but may not have received axitinib.
* Patients must have recovered from any VEGF blocking drug-related toxicity (e.g., proteinuria, hypertension).
* All patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy.
* Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
* Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
* Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
* XRT: At least 14 days after local palliative XRT (small port); At least 150 days must have elapsed if prior TBI, craniospinal XRT or if ≥ 50% radiation of pelvis; At least 42 days must have elapsed if other substantial BM radiation.
* Stem Cell Infusion without TBI: No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant or stem cell infusion.
* Organ Function Requirements
* Adequate Bone Marrow Function Defined As:

  * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)

Adequate Renal Function Defined As:

• Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or

Adequate Liver Function Defined as:

* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
* SGPT (ALT) ≤ 110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
* SGOT (AST) ≤ 125 U/L. For the purpose of this study, the ULN for SGOT is 50 U/L.
* Serum albumin ≥ 2 g/dL.

Adequate Cardiac Function Defined As:

* Shortening fraction of ≥ 27% by echocardiogram, or Ejection fraction of ≥ 50% by gated radionuclide study.
* Must not have a history of myocardial infarction, severe or unstable angina, or peripheral vascular disease.

Adequate Blood Pressure Control Defined As:

A blood pressure (BP) ≤ the 95th percentile for age, height, and gender

Adequate Coagulation Defined As:

* No evidence of active bleeding
* PT and PTT ≤ 1.2 x upper limit of normal (ULN)
* INR ≤1.2

Adequate Pancreatic Function Defined as:

• Lipase ≤ 1.5 x upper limit of normal (ULN).

Exclusion Criteria

* Pregnancy or Breast-Feeding
* Corticosteroids: Patients receiving chronically dosed corticosteroids within 7 days prior to enrollment are not eligible for this trial.
* Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
* Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
* Anti-GVHD agents post-transplant:

Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.

* CYP3A4/5 Inhibitors:

Patients chronically receiving drugs that are known potent CYP3A4/5 inhibitors within 7 days prior to study enrollment, including but not limited to ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit, and grapefruit juice are not eligible

* CYP3A4/5 Inducers:

Patients chronically receiving drugs that are known potent CYP3A4/5 inducers within 7 days prior to study enrollment, including but not limited to rifampin, dexamethasone, phenytoin, carbamazepine, rifabutin, rifapentine, phenobarbital, and St John's wort are not eligible.

* Anti-hypertensives: Patients who are receiving anti-hypertensive medications for control of blood pressure at the time of enrollment are not eligible for this trial.
* Anti-coagulation: Patients who are currently receiving therapeutic anti-coagulation with heparin, low-molecular weight heparin or coumadin are not eligible for this trial.
* Anti-inflammatory or anti-platelet agents: Patients who are currently receiving aspirin, ibuprofen or other non-steroidal anti-inflammatory drugs or anti-platelet agents are not eligible.
* Patients must be able to swallow tablets whole.
* Thyroid Replacement Therapy: Patients who require thyroid replacement therapy are not eligible if they have not been receiving a stable replacement dose for at least 28 days prior to study enrollment. Patients who enter the study on thyroid replacement should have their medication adjusted to maintain TSH in the normal range.

Bleeding and Thrombosis:

Patients with evidence of active bleeding, intratumoral hemorrhage, or bleeding diathesis are not eligible:

* History (within 180 days prior to study enrollment) of arterial thromboembolic events, including transient ischemic attack (TIA) or cerebrovascular accident (CVA).
* History (within 180 days prior to study enrollment) of pulmonary embolism, DVT, or other venous thromboembolic event.
* History of hemoptysis within 42 days prior to study enrollment.

Surgery: Patients who have had or are planning to have the following invasive procedures are not eligible:

* Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment.
* Subcutaneous port placement or central line placement is not considered major surgery but must be placed at least 3 days prior to enrollment for external lines and at least 7 days prior to enrollment for subcutaneous port.
* Core biopsy within 7 days prior to enrollment.
* Fine needle aspirate or central line placement within 7 days prior to enrollment.

CNS disease:

* Patients who have a known primary or metastatic CNS tumor at the time of study enrollment are not eligible. A prior history of metastatic CNS tumor is allowed as long as there is no evidence of CNS disease at study enrollment.
* Patients who have a serious or non-healing wound, ulcer, or bone fracture at the time of study enrollment are not eligible.
* Patients who have a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study enrollment are not eligible.
* Infection: Patients who have known HIV or an uncontrolled infection are not eligible.
* Patients who have received a prior solid organ transplantation are not eligible.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Adverse events as assessed by (CTCAE) version 4.0 | 28 days
MTD of axitinib based on dose-limiting toxicity (DLT) at which fewer than one-third of patients experience DLT, as assessed by CTCAE version 4.0 | 28 days
Pharmacokinetic Assessment of Axitinib Concentrations in Plasma Samples | Day 1 and Day 8 of Cycle 1
  A descriptive analysis of pharmacokinetic (PK) parameters of axitinib will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters.
  Blood samples will be collected at the following time points:Day 1, Cycle 1: Pre-dose, and at 1, 2, 4, 6, and 8 hours after the AM dose on Day 1. Day 8, Cycle 1: Pre-dose, and at 1, 2, 4, 6, and 8 hours after the AM dose on Day 8.

SECONDARY OUTCOMES:
Evaluation of disease response to preliminarily define the antitumor activity of axitinib | up to 2 years
  Patients will have tumor disease evaluations performed at the end of cycles 1, 3, and 5 and then every 3 cycles. Disease response will be assessed according to RECIST criteria for patients with solid tumors and will be reported descriptively. Analyses will be descriptive and exploratory and hypotheses generating in nature.
Biomarkers of kidney injury during axitinib treatment | Cycles 1 and 3
  Proteins in the blood (cystatin C and neutrophil gelatinase-associated lipocalcin (NGAL)) and urine (kidney injury molecule-1 (KIM-1), neutrophil gelatinase-associated lipocalin (NGAL), interleukin-18 (IL-18), creatinine and other markers of renal injury) will be measured before treatment and then weekly during Cycle 1 of axitinib treatment and at the end of Cycle 3

CONTACTS AND LOCATIONS:
Overall Officials: James Geller, MD, Principal Investigator — Children's Oncology Group
Locations (21):
- United States (20):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Childrens Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mark O Hatfield-Warren Grant Magnusun Clinical Center, Bethesda, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Cancer Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada